CLINICAL TRIAL: NCT01631019
Title: Influence of Long-term Cell-phone Based Home Exercise on Biomarkers, Skeletal Muscle and Mortality in Patients With COPD
Brief Title: Mobile-phone-based Home Exercise in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 95-1401B
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-06

CONDITIONS: Moderate to Severe COPD Receiving Home Exercise Training
Keywords: Chronic Obstructive Pulmonary Disease; Pulmonary Rehabilitation; Mobile phone; Biomarker
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- with mobile phone assistance (Active Comparator): In the mobile phone group, patients were asked to continue their exercise program at home at a fixed walking speed. During this period of time, the adherence to protocol was reinforced by telephone from health professionals whenever patients missed one day of their walking training detected by the central system. Patients were asked to continue their exercise program at home at a fixed walking speed, and return to the clinic at 1, 2, 3 and 6 months.
  Interventions: Behavioral: Mobile-phone-based Home Exercise Training Program; Behavioral: Home Exercise Training Program
- with free walk (Placebo Comparator): Patients in the control group were educated the same exercise protocol, but were only verbally asked to freely take the walking exercise training at home. The adherence to the walking exercise at home was reported by the patients themselves at every return visits. All the patients received ISWT, spirometry and blood sample for inflammatory biomarkers at baseline, 1, 2, 3 and 6 months.
  Interventions: Behavioral: Home Exercise Training Program

INTERVENTIONS:
Behavioral: Mobile-phone-based Home Exercise Training Program — Patients in the mobile phone group were asked to perform daily endurance exercise training under mobile phone guidance, and the adherence was reported back to the central server. The level of endurance walking was re-assessed and re-adjusted initially on regular clinical visits every four weeks during the first three months. During this period of time, the adherence to protocol was reinforced by telephone from health professionals whenever patients missed one day of their walking training detected by the central system. Patients were asked to continue their exercise program at home at a fixed walking speed, and return to the clinic at 1, 2, 3 and 6 months.
  Arms: with mobile phone assistance
Behavioral: Home Exercise Training Program — all the subjects were assessed by an incremental shuttle walking test (ISWT) (24) for estimation of exercise endurance. Baseline spirometry and body mass index (BMI) were recorded. The adherence and compliance of the home-based exercise training program was assessed by monitoring the frequency of performance and the duration of the endurance walking program recorded on the central system every week. Patients were asked to continue their exercise program at home at a fixed walking speed, and return to the clinic at 1, 2, 3 and 6 months.

SUMMARY:
Background: Moderate-intensity exercise training improves skeletal muscle aerobic capacity and increased oxidative enzyme activity, as well as exercise tolerance in Chronic Obstructive Pulmonary Disease (COPD) patients.

Design: To investigate the home-based exercise training program can reduce inflammatory biomarkers in COPD.

Setting: Conducted from January 2007 to December 2007 at a tertiary medical center, Chang Gung Memorial Hospital, Taiwan.

Patients: Moderate to severe COPD receiving home exercise training, 12 using mobile phone assistance and 14 with free walk, were assessed for 6 months.

Measurements: Incremental shuttle walk test (ISWT), spirometry, strength of limb muscles, C-reactive protein (CRP) and inflammatory cytokines.

DETAILED DESCRIPTION:
Exercise training is the cornerstone of comprehensive rehabilitation programs in patients with COPD. Exercise training improves skeletal muscle oxidative capacity and efficiency that leads to a less alveolar ventilation at a given work rate. Patients can tolerate a heavier work load with less dyspnea under exercise. To date, it remains unclear whether and to what extent markers of low-grade systemic inflammation may affect trainability in clinically stable patients. Although specific exercise modalities can be applied to reverse muscle dysfunction, exercise intolerance, and reduced health-related quality of life, there is a substantial heterogeneity in the response to exercise training among patients with clinically stable COPD. Endurance exercise training has been reported to have consistently high clinical efficacy. Most pulmonary rehabilitation programs are hospital based and ask patients with regular supervision and monitoring in order to achieve persistent and optimal physiological benefits. However, compliance and time consuming with regular visits to the hospital or clinics are major stumbling blocks to the success of these programs. Recently, the investigators have developed a home-based exercise training program for stable COPD patients by asking them to walk at a speed controlled by the tempo of music from a program installed in a mobile phone. The tempo of music was set to keep the same walking speed at the intended level for endurance exercise training for all patients. Our mobile phone-based system provides an efficient home endurance exercise training program with good compliance and clinical outcomes in patients with moderate-to-severe COPD. This study was therefore designed to further explore whether the circulating level of inflammatory markers, such as CRP, IL-6, TNF-α, and IL-8, will be reduced in patients with COPD undergoing a mobile-phone assisted home-based exercise training program

ELIGIBILITY:
Inclusion Criteria:

* patients with moderate to severe COPD

Exclusion Criteria:

* requirement for oxygen therapy;
* presence of symptomatic cardiovascular diseases or severe systemic diseases limiting exercise capacity;
* use of medications affecting exercise responses;
* musculoskeletal conditions with exercise performance limitation; and
* impaired hearing or vision that affects subject's ability to follow the exercise training program.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
inflammatory cytokines | 6 months
  IL-8
C-reactive protein (CRP) | 6 months
  CRP as systemic inflamatory status
Incremental shuttle walk test (ISWT) | 6 months
  Distence of shuttle walking test!
spirometry | 6 months
  FEV1 and FEV1/FVC.
strength of limb muscles | 6 months
  upper and lower limbs stregth

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan, Taiwan

REFERENCES:
- [Derived] Wang CH, Chou PC, Joa WC, Chen LF, Sheng TF, Ho SC, Lin HC, Huang CD, Chung FT, Chung KF, Kuo HP. Mobile-phone-based home exercise training program decreases systemic inflammation in COPD: a pilot study. BMC Pulm Med. 2014 Aug 30;14:142. doi: 10.1186/1471-2466-14-142. PMID 25175787